CLINICAL TRIAL: NCT06562868
Title: Comparison of the 2-year Clinical Performances of Class II Restorations Using Different Restorative Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevim Hancer Sarica, Research Assistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERU-RDT-SHS-01
Record Dates: First submitted 2024-08-18; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Dental Caries Class II

STUDY DESIGN:
Intervention Model Description: Three groups with different restoration materials
Who Masked: Participant, Outcomes Assessor
Masking Description: While the materials used for the restorations were known to the practitioner, neither the patients nor the specialist dentists conducting the follow-up examinations were aware of them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bulk-fill Composite Resin (Active Comparator): Before starting the restoration procedure, local anesthesia was administered to the tooth or teeth. The caries were removed and the preparation was completed. Following the washing and drying of the cavities, cotton rolls and saliva ejectors were placed to ensure isolation. An appropriate matrix system and wooden wedges were applied. A 0.2% chlorhexidine gluconate solution was used as the cavity disinfectant. Subsequently, the enamel surfaces of the teeth were roughened for 30 seconds using a selective etching technique with 37% phosphoric acid. The universal dental adhesive system was applied according to the manufacturer's instructions. Restorations were performed with Filtek One Bulk Fill Restorative , ensuring that each layer did not exceed 4 mm in thickness.The restorations were evaluated according to FDI criteria at baseline, 1 year and 2 years.
  Interventions: Other: Bulk-fill Composite Resin
- Traditional Posterior Composite Resin (Active Comparator): Before starting the restoration procedure, local anesthesia was administered to the tooth or teeth. The caries were removed and the preparation was completed. Following the washing and drying of the cavities, cotton rolls and saliva ejectors were placed to ensure isolation. An appropriate matrix system and wooden wedges were applied. A 0.2% chlorhexidine gluconate solution was used as the cavity disinfectant. Subsequently, the enamel surfaces of the teeth were roughened for 30 seconds using a selective etching technique with 37% phosphoric acid. The universal dental adhesive system was applied according to the manufacturer's instructions. Restorations were performed with Clearfil Majesty Posterior.The restorations were evaluated according to FDI criteria at baseline, 1 year and 2 years.
  Interventions: Other: Traditional Posterior Composite Resin
- High-filler Flowable Composite Resin (Active Comparator): Before starting the restoration procedure, local anesthesia was administered to the tooth or teeth. The caries were removed and the preparation was completed. Following the washing and drying of the cavities, cotton rolls and saliva ejectors were placed to ensure isolation. An appropriate matrix system and wooden wedges were applied. A 0.2% chlorhexidine gluconate solution was used as the cavity disinfectant. Subsequently, the enamel surfaces of the teeth were roughened for 30 seconds using a selective etching technique with 37% phosphoric acid. The universal dental adhesive system was applied according to the manufacturer's instructions. Restorations were performed with high-filler flowable composite resin.The restorations were evaluated according to FDI criteria at baseline, 1 year and 2 years.
  Interventions: Other: High-filler Flowable Composite

INTERVENTIONS:
Other: Bulk-fill Composite Resin — The evaluation of the restorative material according to FDI criteria at baseline, 1 year and 2 years after application
  Arms: Bulk-fill Composite Resin
Other: Traditional Posterior Composite Resin — The evaluation of the restorative material according to FDI criteria at baseline, 1 year and 2 years after application
  Arms: Traditional Posterior Composite Resin
Other: High-filler Flowable Composite — The evaluation of the restorative material according to FDI criteria at baseline, 1 year and 2 years after application
  Arms: High-filler Flowable Composite Resin

SUMMARY:
The aim of this study is to compare the clinical success of different filling materials used in the treatment of dental caries. Systemically healthy individuals with good oral hygiene and interproximal caries in their posterior teeth participated in the study. Participants underwent initial radiographic and intraoral examinations. Three different filling materials were applied to the participants' teeth. The restorations were evaluated at baseline, 1 year, and 2 years.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the clinical performance of Class II carious defects restored with traditional posterior composite, bulk-fill composite, and high-fill flowable composite resin according to the World Dental Federation (FDI) criteria at 12-month and 24-month intervals. In this study, 110 patients underwent initial radiographic and intraoral examinations. Radiographically, 259 teeth with interproximal caries at D1 and D2 levels were identified. All restorations in the study were performed by the same dentist. Before starting the restoration procedure, local anesthesia was administered to the tooth or teeth. The caries were removed and the preparation was completed. Following the washing and drying of the cavities, cotton rolls and saliva ejectors were placed to ensure isolation. An appropriate matrix system and wooden wedges were applied. A 0.2% chlorhexidine gluconate solution was used as the cavity disinfectant. Subsequently, the enamel surfaces of the teeth were roughened for 30 seconds using a selective etching technique with 37% phosphoric acid. The universal dental adhesive system was applied according to the manufacturer's instructions..The first group received bulk-fill composite resin (Filtek One Bulk Fill Restorative), the second group received traditional posterior composite (Clearfil Majesty Posterior ), and the third group received high-filler flowable composite resin. The same universal dental adhesive system was used for all groups. All restorations were evaluated by two experienced dentists according to the FDI evaluation criteria at baseline,1 year and 2 years. In cases where discrepancies were observed between the two examiners, the assessment was based on a consensus decision made by both dentists. Restorations were evaluated and scored separately for each criterion on a scale from 1 to 5: 1 = clinically excellent, 2 = clinically good, 3 = clinically adequate, 4 = clinically insufficient (requires repair), 5 = clinically poor (requires replacement).

ELIGIBILITY:
Inclusion Criteria:

* The patient has no systemic disease
* The patient should be over 18 years of age
* The patient should have good periodontal status
* Teeth to be restored should be symptomless and vital
* Teeth to be restored should have proximal contacts on both mesial and distal surfaces and be in occlusion with the antagonist teeth
* Teeth that have class II caries lesion in external and middle 1/3 of dentine thickness radiographically

Exclusion Criteria:

* Xerostomia and bruxism
* Absence of adjacent and antagonist teeth
* Extremely poor oral hygiene, severe or chronic periodontitis
* Pregnant or lactating women
* Teeth that have any restoration, endodontic treatment, periodontal and periapical pathology.
* The patients who are undergoing orthodontic treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2024-06-09 (Actual)

PRIMARY OUTCOMES:
FDI World Dental Federation Evaluation Criteria | two years
  The FDI evaluation criteria, developed by the World Dental Federation, are used to assess the clinical performance of dental restorations. The restorations were evaluated separately for each criterion and scored on a scale from 1 to 5: 1 = clinically excellent, 2 = clinically good, 3 = clinically adequate, 4 = clinically insufficient (requires repair), 5 = clinically poor (requires replacement).

CONTACTS AND LOCATIONS:
Overall Officials: Sevim Hancer Sarica, RA, Principal Investigator — Erciyes University Faculty of Dentistry Depertmant of Restorative Dentistry
Locations (1):
- Erciyes University Faculty of Dentistry Department of Restorative Dentistry, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No